CLINICAL TRIAL: NCT04329767
Title: A Prospective Post-Market Study to Evaluate the Clinical Utility of IRIS, a Three-dimensional (3-D) Anatomical Modeling Software for Pre-operative Surgical Planning and Intra-operative Navigation for Nephrectomy
Status: Completed | Type: Observational
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: ISI-IRIS-002
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Kidney Cancer
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- IRIS Arm: Utilize the CT scan along with the IRIS 3D model preoperatively and intraoperatively
  Interventions: Device: IRIS 1.0
- CT Arm: Utilize only the standard 2D CT scan preoperatively and intraoperatively

INTERVENTIONS:
Device: IRIS 1.0 — Intuitive's IRIS 1.0 system is a software only device and service intended to create and deliver segmented image studies (3D anatomical models) based on patients computed tomography (CT) scans. It is intended as software for preoperative surgical planning, and as software for the intraoperative display of the aforementioned multidimensional digital images.
  Groups: IRIS Arm

SUMMARY:
This is a prospective, multi-center, post-market study to evaluate the clinical utility of IRIS, a 3D anatomical modeling software, with standard CT scans during pre-operative planning and intra-operative navigation for nephrectomy. The study will be conducted over the course of 21-24 months and enroll approximately 60-120 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 years or older
2. Subject is undergoing robotic-assisted partial or robotic-assisted radical nephrectomy being performed by participating surgeon
3. Subjects who has had or plan to have a CT scan (with IV contrast medium)

Exclusion Criteria:

1. Subject has a solitary or horseshoe kidney
2. Subject has more than two masses in the applicable kidney requiring multiple partial nephrectomies on the same kidney
3. Subject with prior surgery (ex: partial nephrectomy etc.) on the affected kidney excluding endoscopic kidney stone surgery
4. Subject with renal vein tumor thrombus
5. Subjects planned to have a bilateral operation (ex: bilateral partial nephrectomies planned at the same time)
6. Metastatic disease with life expectancy of less than 1 year
7. Pregnant or suspect pregnancy
8. Subject is mentally handicapped or has a psychological disorder or severe systemic illness that would preclude compliance with study requirements or ability to provide informed consent
9. Subject belonging to other vulnerable population, e.g, prisoner or ward of the state

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with kidney cancer who will undergo robotic-assisted partial or robotic-assisted radical nephrectomy.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Clinical utility of IRIS 3D model with CT scans during Intra-Operative navigation | Intra-operative
  1. Interpretation of the anatomy
  2. Procedure efficiency,
  3. Sufficient information to use intraoperatively, and
  4. Impact on the clinical practice

SECONDARY OUTCOMES:
Clinical utility of IRIS 3D model with CT scans during preoperative surgical planning | Preoperative
  1. Interpretation of the anatomy,
  2. Sufficient information to use preoperatively, and
  3. Confidence in completing the planned procedure.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Hackensack University Medical Center, Edison, New Jersey
  - University of Rochester Medical Center, Rochester, New York